CLINICAL TRIAL: NCT05871398
Title: The Efficacy of Potassium-competitive Acid Blocker (P-CAB) in Patients With Laryngopharyngeal Reflux Disease: a Double- Blind, Randomized, Placebo-controlled Pilot Study
Brief Title: The Efficacy of Potassium-competitive Acid Blocker in Patients With Laryngopharyngeal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-1909-005-096
Record Dates: First submitted 2023-05-02; First posted 2023-05-23 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Laryngopharyngeal Reflux Disease
Keywords: : Laryngopharyngeal reflux disease; potassium-competitive acid blocker; treatment effectiveness
MeSH Terms: interventions — tegoprazan

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- tegoprazan group (Active Comparator)
  Interventions: Drug: Tegoprazan

INTERVENTIONS:
Drug: Tegoprazan — Novel, potent, and highly selective potassium-competitive acid blocker which was developed in Korea
  Arms: tegoprazan group
Drug: Placebo — Placebo
  Arms: placebo group

SUMMARY:
Background/Aims: Tegoprazan is a novel potassium-competitive acid blocker that has a fast onset of action and can control gastric pH for a prolonged period, which could offer clinical benefit in acid-related disorders. The investigators aimed to evaluate whether tegoprazan would be more effective in controlling symptoms than placebo in patients with laryngopharyngeal reflux disease (LPRD). Methods: This double-blind, randomized, placebo-controlled trial randomly assigned 35 patients suffering LPRD symptom to two groups: Tegoprazan50mg once daily and placebo. The primary end point was complete resolution rate of LPRD symptoms after 8-week medication, and the secondary endpoints were complete resolution rate of LPRD symptoms after 4-week medication, change of reflux symptom index (RSI) and reflux finding score (RFS) from baseline at 4- and 8-week medication.

ELIGIBILITY:
Inclusion Criteria:

* At least one symptom of LPRD (hoarseness, globus, persistent throat discomfort, and frequent throat clearing) for at least 4 weeks
* Reflux symptom index > 13 and reflux finding score ≥ 7

Exclusion Criteria:

* Viral or bacterial laryngopharyngitis at present
* History of malignancy of head and neck region, esophagus and stomach
* Previous radiotherapy or endotracheal intubation within three months
* Previous anti-reflux surgery or gastroesophageal surgery
* Diagnosis of depression, anxiety, panic, somatoform or other psychotic disorder
* Taking anti-psychotics, anti-depressants or anti-anxiety drugs
* Anti-reflux medication such as proton-pump inhibitors (within 4 weeks before screening), histamine receptor 2 blockers, antacids or prokinetics (within 2 weeks before screening)
* Need for continuous therapy with non-steroidal anti-inflammatory drugs
* Pregnant or breastfeeding women, as well as female patients who were not willing to use contraception for the duration of the clinical trial period
* Abnormal laboratory test values at screening (blood urea nitrogen and serum creatine level >1.5 upper limit of normal [ULN]; total bilirubin levels and serum levels of alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and gamma-glutamyl transferase > 2 ULN) or
* Any other conditions or disease that an investigator considered not appropriate for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Reflux symptom index (RSI) | Week 8
  RSI is a validated nine-item, self-administered questionnaire to assess the severity and responses to treatment of laryngopharyngeal reflux disease-associated symptoms. Each component is scored between 0 (no problem) and 5 (severe problem), with a maximum total score of 45.
  Non-response = RSI ≥ 13, Response = post-treatment RSI < 13 and change in RSI < 50%, Complete response = post-treatment RSI < 13 and change in RSI ≥ 50%.
Reflux finding score (RFS) | Week 8
  RFS is a validated rating scale developed to quantify the degree of laryngeal involvement in laryngopharyngeal reflux disease during fiberoptic laryngoscopy. Scores range from 0 (no abnormal findings) to 26 (worst score possible).
  Normal < 7, Abnormal ≥ 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Pusan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lechien JR, Saussez S, Karkos PD. Laryngopharyngeal reflux disease: clinical presentation, diagnosis and therapeutic challenges in 2018. Curr Opin Otolaryngol Head Neck Surg. 2018 Dec;26(6):392-402. doi: 10.1097/MOO.0000000000000486. PMID 30234664
- [Background] Katzka DA, Kahrilas PJ. Advances in the diagnosis and management of gastroesophageal reflux disease. BMJ. 2020 Nov 23;371:m3786. doi: 10.1136/bmj.m3786. PMID 33229333
- [Derived] Jeon HK, Kim GH, Cheon YI, Shin SC, Lee BJ. Efficacy of Tegoprazan in Patients with Laryngopharyngeal Reflux Disease: A Preliminary Feasibility Study. J Clin Med. 2023 Sep 22;12(19):6116. doi: 10.3390/jcm12196116. PMID 37834761